CLINICAL TRIAL: NCT05235893
Title: The Effect of Reflexology on Pain Management in Newborns: A Randomized-Controlled Clinical Study
Brief Title: Effect of Reflexology on Pain Management in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, mahmut caner us, Medical Doctor, PhD student, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019/406
Record Dates: First submitted 2021-11-17; First posted 2022-02-11 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Pain, Procedural; Pain, Acute; Analgesia
Keywords: newborn; pain management; crying; analgesics; reflexology
MeSH Terms: conditions — Pain, Procedural; Acute Pain; Agnosia; Crying | interventions — Musculoskeletal Manipulations; Kangaroo-Mother Care Method; Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Reflexology Group (Experimental): The newborns who have applied Reflexology to soles three minutes before and during 5-7 minutes of painful procedure by a physiotherapist, certificated in reflexology.
  Interventions: Procedure: Reflexology
- Sucrose Group (Active Comparator): The newborns who were given one ml of a single-use 24% concentration of sucrose solution in the form of ready to use preparations
  Interventions: Procedure: Sucrose %24
- Kangaroo Care Group (Active Comparator): The newborns who were placed on the mother's lap for 3-5 minutes before the painful intervention and kangaroo care was applied
  Interventions: Procedure: Kangaroo care
- Music Group (Active Comparator): Newborns who were exposed to the recorded "Deep Sleep" track from "Bedtime Mozart: Classical Lullabies for Babies" music
  Interventions: Procedure: Music
- Control Group (No Intervention): Control arm

INTERVENTIONS:
Procedure: Reflexology — Reflexology was applied to soles of the babies in the second study group during 5-7 minutes, three minutes before the painful procedure was started by a physiotherapist, certificated in reflexology.
  Arms: Reflexology Group
Procedure: Sucrose %24 — The newborns who were given one ml of a single-use 24% concentration of sucrose solution in the form of ready to use preparations
  Arms: Sucrose Group
Procedure: Kangaroo care — The newborns who were placed on the mother's lap for 3-5 minutes before the painful intervention and kangaroo care was applied
  Arms: Kangaroo Care Group
Procedure: Music — Newborns who were exposed to the recorded "Deep Sleep" track from "Bedtime Mozart: Classical Lullabies for Babies" music
  Arms: Music Group

SUMMARY:
Introduction: Approximately 10-14 painful procedures per day are performed in preterm and term infants during the hospital stay in the first week. The investigators aimed to determine the effect of reflexology being applied to the sole during painful procedures on pain perception, behavioral responses, and physiological changes in newborns compared with other non-pharmacological methods.

Material and Method: This study was planned as a randomized controlled trial in term infants being followed up in the Neonatal Intensive Care Unit (NICU) and maternity ward. To reduce pain during attempts to collect venous blood or heel lance which are routinely applied to term newborns before discharge; reflexology on the soles of the foot, 24% sucrose solution, kangaroo care, listening to classical music were applied to the babies and were compared to those who did not have any analgesic method.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled trial conducted between December 2019 and March 2020 in term babies being followed up in the NICU and maternity ward. To reduce pain during attempts to collect venous blood or heel lance which are routinely applied to term newborns before discharge; reflexology on the soles of the foot, 24% sucrose solution, kangaroo care, listening to classical music were applied to the babies and were compared to those who have not applied any analgesic method. All term infants were collected by the convenience sampling method from NICU and maternity ward according to inclusion and exclusion criteria. The parents of all participants were informed in detail about the study by investigator 1, and a copy of the informed consent form was delivered to the family. During the study period (December 2019 and March 2020), an average of 915 neonates per month was born in the same hospital. The participants who met the selection criteria and whose mothers agreed to participate in the study were recruited. A computer-generated block method assigned infants to receive either reflexology, 24% sucrose, kangaroo care, classic music, or control group. Term newborns hospitalized in the maternity ward and the NICU are randomly allocated to one of five groups, before the heel stick procedure by investigator 1 using a computer-generated table. For each participant, a random number was generated, and babies were subgrouped as follows: 1) Sucrose Group, 2) Reflexology Group, 3) Kangaroo Care Group, 4) Music Group, 5) Control Group, and the same randomization method was used to allocate the newborns before venous sampling. Sampling size was calculated as 27 per group and total number as 270 to obtain statistical significance with at least 85% power, and for an alpha significance level of 0.05 respectively in five groups. 30 newborns were allocated to each group for venous sampling (Total 150) and heel-prick (Total 150) intervention taking into account drop-out and other possible problems.

Interventions One ml of a single-use 24% concentration of sucrose solution in the form of ready-to-use preparations were given to the newborns in the first study group by the investigator 2, two minutes before the painful intervention. Reflexology was applied to soles of the babies in the second study group during 5-7 minutes, three minutes before the painful procedure was started by a physiotherapist, certificated in reflexology. The participants in the third study group were placed on the mother's lap for 3-5 minutes before the painful intervention and kangaroo care was applied. Participants in the fourth study group were exposed to the recorded music with sounds up to 60 A-weighted decibels, starting 20 minutes before the intervention, continuing for 7 minutes after the procedure. Music was administered using the "Deep Sleep" track from "Bedtime Mozart: Classical Lullabies for Babies" (2011), an instrumental lullaby music track chosen after discussion with a music therapist for stability, repeatability, and presence of minor tones. The piece of music was presented as a loop and was played back from a sound source using 2 high-quality portable speakers, placed equidistant from the head on each side. The sound levels at both ears were checked after speaker placement and the sound was gradually scaled up to the study limit of 60 A-weighted decibels. However, the total auditory exposure was checked to ensure that it remained within the recommended limits at the ear level.

Sampling procedures Heel pricks and venous blood collection were performed by an experienced nurse blinded to the applied non-pharmacological analgesic method (heel lance by nurse 1 / venous sampling by nurse 2). BD Quickheel Preemie lancet; Becton, Dickinson and Company, East Rutherford, NJ was used for heel lance. The blood-drawing procedure was conducted by an experienced newborn nurse in one attempt and the same amount of blood was taken from each newborn. The blood drawing site was the lateral surface of the right heel. During the data collection process, parents could observe their newborns in both the study and control groups. All interventions were made after all infants were followed up in the prone or side-lying position, feeding, and then cleaned in the NICU or maternity ward.

Pain Assessment Pain assessments, physiological and behavioral responses of participants were measured during the interventions. Behavioral responses and pain assessments of all newborn infants were evaluated with Neonatal Infant Pain Scale (NIPS) by 2 different investigator (3-4) before (2 minutes ago), during and after (after 2 minutes) interventions, and physiological changes were recorded by pulse oximetry (the Masimo Rad 5 Pulse Oximeter, Masimo Corporation, Irvine, CA). NIPS and other data were filled via video recordings by experienced NICU nurses and forms were sent by mail to the department to be analyzed, separately. NIPS was developed by Lawrence et al in 1993 to assess behavioral responses and physiologic pain responses of preterm and full-term newborns during acute pain and was adapted to the Turkish version by Akdovan in 1999. Lawrence et al. found the reliability coefficient of NIPS to be in the range of .92-.97. In addition, Akdovan reported the Cronbach's value to be between .83 and .86 in the Turkish version. The scale comprised five behavioral indicators (facial expressions, cry, state of arousal, arms, legs) and one physiologic indicator (breathing patterns). Except for ''cry,'' which had three possible score descriptors (0, 1, or 2), each behavioral indicator was scored with 0 or 1. The total score ranged between 0 and 7. High scores indicated higher levels of pain. An oximeter was secured to the participants before the intervention and peak heart rates and oxygen saturation values were obtained. The probe of the pulse oximeter was attached to the left foot of the newborns and was fixed so that it would remain in place. Heartbeat (HR), respiratory rate (RR), body temperature (BT), blood pressure (systolic blood pressure (BPs), diastolic blood pressure (DBp), mean arterial pressure (MAP), oxygen saturation (SpO2) values were recorded on the follow-up form.

Ethical approval: The study was approved by the ethics committee of the Local Health District with decision number: 2019-25-02 at 23.12.2019. Informed written consent was obtained from the parents before recruitment.

Statical Analysis Statistical Package for the Social Sciences (SPSS 15.0) for Windows program was used for statistical analysis. Descriptive statistics; number and percentage for categorical variables, and numerical variables as mean, standard deviation, minimum, maximum, median. Since the numerical variables did not meet the normal distribution condition, comparisons of two independent groups were made with the Mann-Whitney U Test. Since the differences of numerical variables in the dependent groups did not meet the normal distribution condition, they were compared with the Wilcoxon test. Inter-rater reliability bias was evaluated with the Intraclass Correlations (ICC) level. Bonferroni's correction was used to evaluate inter-method efficacy and a one-way ANOVA test was used to investigate more than 2 independent variables. Statistical alpha significance level was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Newborns who are hospitalized in the NICU and maternity ward who will undergo heel lance or venous blood sampling before discharge.
* Those who meet the discharge criteria recommended in the TNS guideline
* Approved family informed consent.

Exclusion Criteria:

* Infants born with a birth weight below 2500 g and over 4000 g
* Infants born before 37 gestational weeks,
* Presence of major congenital anomaly or neurological problems.

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Effect of Reflexology on change in pain perception during painful procedures in Newborns | 2 minutes before (pre-intervention), at the beginning of the intervention, and 2 minutes after (immediately after the intervention) the painful interventions
  To evaluate the effect of reflexology on pain perception, Neonatal Infant Pain Scale was scored and compared with other non-pharmacological methods outcomes. Scoring was obtained 2 minutes before, during, and 2 minutes after the painful intervention in babies aged 2 to 28 days, before discharge from hospital. The Neonatal Infant Pain Scale consists of five behavioral sections and one physiological section including facial expression, crying, breathing, arm, and leg movements, and alertness. Total scores for each section range between 0 and 7. Scores from 0 to 2 indicate mild to no pain, 3 to 4 indicate mild to moderate pain, and > 4 indicates severe pain. Higher scores indicate more severe pain. Change from Baseline of Neonatal Infant Pain Scale score was assesed.
Effect of Reflexology on crying time during painful procedures in Newborns | from beginning of the painful intervention until crying stops measured in minutes
  To evaluate the effect of reflexology on behavioural responses, crying time (minute) was noted and compared with other non-pharmacological methods outcomes. During the painful procedures in babies aged 2 to 28 days, crying time was observed by using a chronometer and noted as minutes and seconds. Higher minutes indicate more severe pain.
Effect of Reflexology on change in blood pressure during painful procedures in Newborns | 2 minutes before (pre-intervention), at the beginning of the intervention, and 2 minutes after (immediately after the intervention) the painful interventions
  To evaluate the effect of reflexology on physiological parameters a monitor was used to measure blood pressure (systolic, diastolic, mean arterial pressure; mmHg) and compared with other nonpharmacological methods outcomes. Measurements were obtained 2 minutes before, during, and 2 minutes after the painful intervention in babies aged 2 to 28 days, before discharge from the hospital. Change from the Baseline of blood pressure (systolic, diastolic, mean arterial pressure; mmHg) were assessed.
Effect of Reflexology on change in oxygen saturation during painful procedures in Newborns | 2 minutes before (pre-intervention), at the beginning of the intervention, and 2 minutes after (immediately after the intervention) the painful interventions
  To evaluate the effect of reflexology on physiological parameters a monitor was used to oxygen saturation (%), and compared with other nonpharmacological methods outcomes. Measurements were obtained 2 minutes before, during, and 2 minutes after the painful intervention in babies aged 2 to 28 days, before discharge from the hospital. Change from the Baseline of oxygen saturation (%) was assessed.

SECONDARY OUTCOMES:
Effect of Reflexology on change in heart rate during painful procedures in Newborns | 2 minutes before (pre-intervention), at the beginning of the intervention, and 2 minutes after (immediately after the intervention) the painful interventions
  To evaluate the effect of reflexology on physiological parameters a monitor was used to measure heart rate (/minute) and compared with other nonpharmacological methods outcomes. Measurements were obtained 2 minutes before, during, and 2 minutes after the painful intervention in babies aged 2 to 28 days, before discharge from the hospital. Change from Baseline of heart rate (/minute) was assessed
Effect of Reflexology on change in respiratory rate during painful procedures in Newborns | 2 minutes before (pre-intervention), at the beginning of the intervention, and 2 minutes after (immediately after the intervention) the painful interventions
  To evaluate the effect of reflexology on physiological parameters a monitor was used to measure respiratory rate (/minute) and compared with other nonpharmacological methods outcomes. Measurements were obtained 2 minutes before, during, and 2 minutes after the painful intervention in babies aged 2 to 28 days, before discharge from the hospital. Change from Baseline of respiratory rate (/minute) was assessed

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Caner US, MD, Principal Investigator — Esenler Maternity and Child Health Hospital
Locations (1):
- Esenler Maternity and Child Health Hospital, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Provided that patient information is kept confidential, it will only be shared with the consent of the families when evaluated and deemed appropriate by the researchers.

REFERENCES:
- [Background] Huang RR, Xie RH, Wen SW, Chen SL, She Q, Liu YN, Harrison D. Sweet Solutions for Analgesia in Neonates in China: A Systematic Review and Meta-Analysis. Can J Nurs Res. 2019 Jun;51(2):116-127. doi: 10.1177/0844562118803756. Epub 2018 Nov 22. PMID 30466313
- [Background] Benoit B, Martin-Misener R, Latimer M, Campbell-Yeo M. Breast-Feeding Analgesia in Infants: An Update on the Current State of Evidence. J Perinat Neonatal Nurs. 2017 Apr/Jun;31(2):145-159. doi: 10.1097/JPN.0000000000000253. PMID 28437305
- [Background] Hall RW, Anand KJ. Pain management in newborns. Clin Perinatol. 2014 Dec;41(4):895-924. doi: 10.1016/j.clp.2014.08.010. Epub 2014 Oct 7. PMID 25459780
- [Background] Yilmaz D, Yilmaz Kurt F. The effect of foot reflexology on procedural pain before heel lancing in neonates. Arch Pediatr. 2021 May;28(4):278-284. doi: 10.1016/j.arcped.2021.02.015. Epub 2021 Mar 11. PMID 33715931
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Background] Kulkarni A, Kaushik JS, Gupta P, Sharma H, Agrawal RK. Massage and touch therapy in neonates: the current evidence. Indian Pediatr. 2010 Sep;47(9):771-6. PMID 21048258
- [Derived] Us MC, Saran MG, Cebeci B, Akkus E, Seker E, Aybar SSS. A Randomized Comparative Effectiveness Study of Reflexology, Sucrose, and Other Treatments for Needle Procedures in Newborns. Pediatr Neurol. 2023 Mar;140:78-85. doi: 10.1016/j.pediatrneurol.2022.11.019. Epub 2022 Dec 5. PMID 36608413